CLINICAL TRIAL: NCT03315520
Title: A Phase II, Multicenter, Prospective, Non-randomised, Open-label, Clinical Trial to Evaluate Effectiveness and Safety of BeEAC Conditioning Regimen in Malignant Lymphoma Subjects With Indications to Autologous Hematopoietic Stem-cell Transplantation
Brief Title: BeEAC Conditioning Regimen in Malignant Lymphoma Subjects With Indications to Autologous Hematopoietic Stem-cell Transplantation
Acronym: BeEAC-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeEAC-1
Record Dates: First submitted 2017-09-26; First posted 2017-10-20 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Relapsed/Refractory Malignant Lymphomas
Keywords: Hodgkin Lymphoma; Non-Hodgkin lymphoma; autologous hematopoietic stem-cell transplantation; conditioning regimen
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Cytarabine; Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/refractory malignant lymphomas (Experimental): Malignant Lymphoma Subjects With Indications to Autologous Hematopoietic Stem-cell Transplantation using BeEAC (Bendamustine, Cytarabine, Etoposide, Cyclophosphamide) conditioning regimen
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — BeEAC conditioning regimen:
  bendamustine 200 mg/м2 D-6 - D-5; cytarabine 400 mg/м2 D-4 - D-1; etoposide 400 mg/м2 D-4 - D-1; cyclophosphamide 140 mg/м2 totally, divided in 4 days (D-4 - D-1)
  Other Names: Cytarabine; Etoposide; Cyclophosphamide

SUMMARY:
Nowadays there is no randomized trials for comparison the effectiveness and tolerability of different conditioning regimens.

Bendamustine is a unique chemotherapeutic agent that combines alkylating action of nitrogen mustard and the activity of purine antimetabolite. Bendamustine has shown its effectiveness for the treatment of patients with chronic lymphoproliferative diseases such as chronic lymphocytic leukemia and several indolent lymphomas. The literature also presents evidence of the effectiveness bendamustine in patients with Hodgkin's lymphoma who received multiple lines of prior chemotherapy, including high dose chemotherapy and transplantation of peripheral hematopoietic stem cells. There are also data of using bendamustine as a part of conditioning regimen.

In this context, it was planned a study for evaluation the safety and effectiveness of the BeEAC (bendamustine, etoposide, cytarabine, cyclophosphamide) conditioning regimen prior to autologous transplantation of peripheral hematopoietic stem cells for the treatment of relapsed/refractory malignant lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial
2. Be ≥ 18 years of age on day of signing informed consent
3. Eastern Cooperative Oncology Group (ECOG) < 2.
4. Relapsed/refractory malignant lymphoma patients with indications to autologous hematopoietic stem-cell transplantation

Exclusion Criteria:

1. Participation in another clinical trials
2. Clinically relevant heart disease:

   * Myocardial infarction during previous 6 months
   * Unstable angina during previous 3 months
   * Congestive heart failure (III-IV NYHA)
   * Clinically relevant ventricular arrhythmias
   * corrected QT interval (QTc) > 460 мс on ECG (calculated using Frederics formula)
   * Left ventricular ejection fraction ≤ 45% on Echocardiogram
   * Atrial Hypotension (systolic pressure < 86 mmHg) or bradycardia (< 50 per minute, exclusion - drug-induced bradycardia)
   * Uncontrolled arterial hypertension (systolic pressure > 170 mmHg or diastolic pressure > 105 mmHg)
3. Severe renal dysfunction (serum creatinine > 250 µmol/l)
4. Severe hepatic dysfunction (total bilirubin > 40 µmol/l)
5. Known history of Human Immunodeficiency Virus or active Hepatitis B and C
6. Psychiatric or substance abuse disorders that would interfere with the cooperation with the requirements of the trial
7. Hypersensitivity to investigational drugs
8. Pregnant or breastfeeding females or males and females with childbearing potential must be willing to use an adequate method of birth control (intrauterine device, vasectomy of female subjects' male partner, contraceptive rod implanted into the skin, combination method - (requires use of two of the following) diaphragm with spermicide, cervical cap spermicide, contraceptive sponge, condom, hormonal contraceptive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From admission till discharge from the hospital (approximately 30 days)
  The primary safety analysis will be based on subjects who experienced toxicities as defined by CTCAE criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received BeEAC including serious adverse events (SAEs).
  Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE 4.03. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading and action taking with regard to trial treatment (Incidence of Treatment-Emergent Adverse Events).

SECONDARY OUTCOMES:
Overall Survival | 2 years
Progression-Free Survival | 2 years
Retrospective Comparison of Overall Survival between Carmustine, Etoposide, Cytarabine, Melphalan (BEAM), Cyclophosphamide, Carmustine, Etoposide(CBV) and BeEAC conditioning regimens | 2 years
  The analysis will be based on comparison of overall survival between different conditioning regimens
Retrospective Comparison of Progression-Free Survival between Carmustine, Etoposide, Cytarabine, Melphalan (BEAM), Cyclophosphamide, Carmustine, Etoposide(CBV) and BeEAC conditioning regimens | 2 years
  The analysis will be based on comparison of Progression-Free survival between different conditioning regimens

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav Sarzhevskiy, MD, PhD, Principal Investigator
Locations (1):
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martino M, Olivieri A, Offidani M, Vigna E, Moscato T, Fedele R, Montanari M, Console G, Gentile M, Messina G, Irrera G, Morabito F. Addressing the questions of tomorrow: melphalan and new combinations as conditioning regimens before autologous hematopoietic progenitor cell transplantation in multiple myeloma. Expert Opin Investig Drugs. 2013 May;22(5):619-34. doi: 10.1517/13543784.2013.788643. Epub 2013 Apr 4. PMID 23550793
- [Background] Schmitz N, Pfistner B, Sextro M, Sieber M, Carella AM, Haenel M, Boissevain F, Zschaber R, Muller P, Kirchner H, Lohri A, Decker S, Koch B, Hasenclever D, Goldstone AH, Diehl V; German Hodgkin's Lymphoma Study Group; Lymphoma Working Party of the European Group for Blood and Marrow Transplantation. Aggressive conventional chemotherapy compared with high-dose chemotherapy with autologous haemopoietic stem-cell transplantation for relapsed chemosensitive Hodgkin's disease: a randomised trial. Lancet. 2002 Jun 15;359(9323):2065-71. doi: 10.1016/S0140-6736(02)08938-9. PMID 12086759
- [Background] Blay J, Gomez F, Sebban C, Bachelot T, Biron P, Guglielmi C, Hagenbeek A, Somers R, Chauvin F, Philip T. The International Prognostic Index correlates to survival in patients with aggressive lymphoma in relapse: analysis of the PARMA trial. Parma Group. Blood. 1998 Nov 15;92(10):3562-8. PMID 9808548
- [Background] Chen YB, Lane AA, Logan B, Zhu X, Akpek G, Aljurf M, Artz A, Bredeson CN, Cooke KR, Ho VT, Lazarus HM, Olsson R, Saber W, McCarthy P, Pasquini MC. Impact of conditioning regimen on outcomes for patients with lymphoma undergoing high-dose therapy with autologous hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2015 Jun;21(6):1046-1053. doi: 10.1016/j.bbmt.2015.02.005. Epub 2015 Feb 14. PMID 25687795
- [Background] Friedberg JW, Cohen P, Chen L, Robinson KS, Forero-Torres A, La Casce AS, Fayad LE, Bessudo A, Camacho ES, Williams ME, van der Jagt RH, Oliver JW, Cheson BD. Bendamustine in patients with rituximab-refractory indolent and transformed non-Hodgkin's lymphoma: results from a phase II multicenter, single-agent study. J Clin Oncol. 2008 Jan 10;26(2):204-10. doi: 10.1200/JCO.2007.12.5070. Erratum In: J Clin Oncol. 2008 Apr 10;26(11) 1911. PMID 18182663
- [Background] Knauf WU, Lissitchkov T, Aldaoud A, Liberati AM, Loscertales J, Herbrecht R, Juliusson G, Postner G, Gercheva L, Goranov S, Becker M, Fricke HJ, Huguet F, Del Giudice I, Klein P, Merkle K, Montillo M. Bendamustine compared with chlorambucil in previously untreated patients with chronic lymphocytic leukaemia: updated results of a randomized phase III trial. Br J Haematol. 2012 Oct;159(1):67-77. doi: 10.1111/bjh.12000. Epub 2012 Aug 4. PMID 22861163
- [Background] Moskowitz AJ, Hamlin PA Jr, Perales MA, Gerecitano J, Horwitz SM, Matasar MJ, Noy A, Palomba ML, Portlock CS, Straus DJ, Graustein T, Zelenetz AD, Moskowitz CH. Phase II study of bendamustine in relapsed and refractory Hodgkin lymphoma. J Clin Oncol. 2013 Feb 1;31(4):456-60. doi: 10.1200/JCO.2012.45.3308. Epub 2012 Dec 17. PMID 23248254
- [Background] Visani G, Malerba L, Stefani PM, Capria S, Galieni P, Gaudio F, Specchia G, Meloni G, Gherlinzoni F, Giardini C, Falcioni S, Cuberli F, Gobbi M, Sarina B, Santoro A, Ferrara F, Rocchi M, Ocio EM, Caballero MD, Isidori A. BeEAM (bendamustine, etoposide, cytarabine, melphalan) before autologous stem cell transplantation is safe and effective for resistant/relapsed lymphoma patients. Blood. 2011 Sep 22;118(12):3419-25. doi: 10.1182/blood-2011-04-351924. Epub 2011 Aug 3. PMID 21816830